CLINICAL TRIAL: NCT01382303
Title: Effect of Pentoxifylline on Proteinuria in Korean Type 2 Diabetic Patients : Prospective, Randomized, Double Blinded Active Control, Multicenter Study
Brief Title: Effect of Pentoxifylline on Proteinuria in Korean Type 2 Diabetic Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ajou University School of Medicine (Other)
Collaborators: Bundang CHA Hospital (Other); Hallym University Medical Center (Other); Gangnam Severance Hospital (Other); Yonsei University (Other); Myongji Hospital (Other)
Responsible Party: Principal Investigator, Kwan Woo Lee, professor, Ajou University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AJIRB-MED-CT4-10-055
Record Dates: First submitted 2011-06-22; First posted 2011-06-27 (Estimated); Results first posted 2017-06-16 (Actual); Last update posted 2017-06-16 (Actual); Status verified 2017-03

CONDITIONS: Type 2 Diabetes
Keywords: Type 2 Diabetes; pentoxifylline; proteinuria
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Proteinuria | interventions — Pentoxifylline

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Pentoxifylline (Active Comparator): Pentoxifylline 400mg three times a day
  Interventions: Drug: Pentoxifylline
- Placebo (Placebo Comparator): placebo tablet
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Pentoxifylline — Pentoxifylline 400mg three times a day
  Other Names: Trental
  Arms: Pentoxifylline
Drug: Placebo — placebo tablet three times a day
  Arms: Placebo

SUMMARY:
This multi-center, randomized controlled study aims to evaluate the effects of pentoxifylline on proteinuria in Korean type 2 diabetic patients.

DETAILED DESCRIPTION:
The investigators will recruit adults patients with type 2 diabetes aged over 20 years with spot urine albumin to creatinine ratio over 30mg/g in two consecutive measurements.

Enrolled patients will be randomly assigned to receive pentoxifylline (400mg three times daily) or placebo for 24 weeks.

Fasting blood and spot urine will be collected at baseline, 12 weeks and 24 weeks.

The investigators will evaluate the impact of pentoxifylline on proteinuria in type 2 diabetic patients.

ELIGIBILITY:
Inclusion Criteria:

* type 2 diabetes mellitus
* age >=20 years
* spot urine albumin/creatinine ratio > 30mg/g in two consecutive measurements
* patients on ACE-inhibitor or ARB as an anti-hypertensive drug
* blood pressure <= 150/100 mmHg
* HbA1c <10%

Exclusion Criteria:

* taking insulin pentoxifylline, cilostazol, ketas, viagra in 3 months
* ischemic heart disease, stroke, malignant disease, severe infection in 6 months
* serum creatinine > 2.0mg/dl
* severe liver disease or AST, ALT > 3* ULM
* taking systemic steroid in 1 month
* pregnant or plan to become pregnant during the clinical trial
* lactation

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 174 (Actual)
Dates: Start 2010-10-25 (Actual); Primary Completion 2013-12-20 (Actual); Study Completion 2013-12-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kwan-Woo Lee, PhD, Principal Investigator — Ajou University School of Medicine
Locations (1):
- Ajou University Hospital, Suwon, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Colombijn JM, Hooft L, Jun M, Webster AC, Bots ML, Verhaar MC, Vernooij RW. Antioxidants for adults with chronic kidney disease. Cochrane Database Syst Rev. 2023 Nov 2;11(11):CD008176. doi: 10.1002/14651858.CD008176.pub3. PMID 37916745
- [Derived] Han SJ, Kim HJ, Kim DJ, Sheen SS, Chung CH, Ahn CW, Kim SH, Cho YW, Park SW, Kim SK, Kim CS, Kim KW, Lee KW. Effects of pentoxifylline on proteinuria and glucose control in patients with type 2 diabetes: a prospective randomized double-blind multicenter study. Diabetol Metab Syndr. 2015 Jul 19;7:64. doi: 10.1186/s13098-015-0060-1. eCollection 2015. PMID 26300986

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Pentoxifylline | Placebo
Started | 87 | 87
Completed | 52 | 70
Not Completed | 35 | 17

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Pentoxifylline | Placebo | Total
Number analyzed (Participants) | 87 | 87 | 174
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.7 (10.1) | 63.8 (9.4) | 63.8 (9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 40 | 31 | 71
  Male | 47 | 56 | 103
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Korea, Republic of | 87 | 87 | 174

OUTCOME MEASURES:

1. Primary Outcome: Percentage Change in Proteinuia
Description: Changes of urine protein to creatinie ratio from baseline to 24 weeks
Time Frame: baseline and 24 weeks
Measure: Mean (Inter-Quartile Range); unit: % change from baseline
Arm/Group | Pentoxifylline | Placebo
Number analyzed (Participants) | 52 | 70
% change from baseline | -23 [-50 to 10] | -4 [-30 to 40]

2. Secondary Outcome: Percentage Change in Albuminuria
Description: Changes of urine albumin to creatinie ratio from baseline to 24 weeks
Time Frame: baseline and 24 weeks
Measure: Mean (Inter-Quartile Range); unit: % change from baseline
Arm/Group | Pentoxifylline | Placebo
Number analyzed (Participants) | 52 | 70
% change from baseline | -10 [-47 to 50] | -6 [-45 to 41]

3. Secondary Outcome: Mean Change of eGFR
Description: changes in eGFR from baseline to 24 weeks
Time Frame: baseline and 24 weeks
Measure: Mean (Standard Deviation); unit: ml/min per 1.73m2
Arm/Group | Pentoxifylline | Placebo
Number analyzed (Participants) | 52 | 70
ml/min per 1.73m2 | -1.05 (18.20) | -3.59 (14.20)

4. Secondary Outcome: Mean Change of Creatinine
Description: changes serum creatinine from baseline to 24 weeks
Time Frame: baseline and 24 weeks
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Pentoxifylline | Placebo
Number analyzed (Participants) | 52 | 70
mg/dL | 0.03 (0.16) | 0.04 (0.15)

5. Secondary Outcome: Mean Change of Fasting Glucose
Description: changes serum fasting glucose from baseline to 24 weeks
Time Frame: baseline and 24 weeks
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Pentoxifylline | Placebo
Number analyzed (Participants) | 52 | 70
mg/dL | -10.0 (38.9) | 8.4 (37.4)

6. Secondary Outcome: Mean Change of TNF-a
Description: changes in TNF-a from baseline to 24 weeks
Time Frame: baseline and 24 weeks
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Pentoxifylline | Placebo
Number analyzed (Participants) | 52 | 70
pg/mL | -0.24 (3.11) | 0.14 (0.71)

ADVERSE EVENTS:
Arm/Group | Pentoxifylline | Placebo
Serious Adverse Events (participants affected / at risk) | 0/87 | 0/87
Other Adverse Events (participants affected / at risk) | 20/87 | 3/87
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Pentoxifylline (N=87) | Placebo (N=87)
dyspepsia (Gastrointestinal disorders) | 7 | 1
nasea (Gastrointestinal disorders) | 5 | 2
gastric reflux (Gastrointestinal disorders) | 5 | 3
headache (Vascular disorders) | 3 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No